CLINICAL TRIAL: NCT00189241
Title: An Open-Label Study to Evaluate the Safety and Long-Term Clinical Efficacy of Imiquimod 5% Cream Applied Once Daily 5 Days Per Week for 6 Weeks in the Treatment of Superficial Basal Cell Carcinoma
Brief Title: A Study to Evaluate Effectiveness of Imiquimod 5% Cream in Superficial Basal Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Organization: Viatris Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1412-IMIQ
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2010-08

CONDITIONS: Basal Cell Carcinoma
Keywords: Aldara; Superficial Basal Cell Carcinoma; Long-Term Study
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Imiquimod

INTERVENTIONS:
Drug: imiquimod

SUMMARY:
The purpose of this study is to evaluate the long-term sustained clearance rate of superficial basal cell carcinoma during a 5 year period following treatment with imiquimod

ELIGIBILITY:
Inclusion Criteria:

* Have one superficial BCC - primary tumour
* Minimum tumour area of 0.5cm2, maximum diameter of 2.0cm.
* If female and of child bearing potential, negative pregnancy test and willing to use medically acceptable method of contraception.

Exclusion Criteria:

* Evidence of clinically significant, unstable medical conditions.
* Evidence of Gorlin syndrome, metastatic tumour or tumour with high probability of metastatic spread, have or have had within last 5 years other malignant cancers of the skin at target tumour site.
* Have received defined treatments in tumour site or surrounding area.
* Any dermatological disease in the target tumour site or surrounding area.
* Have had a systemic bacterial or viral infection within 2 weeks prior to study initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2001-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the long-term sustained clearance rate, defined as the proportion of subjects who are clinically clear of sBCC at the treated sBCC target tumour site at the 12 week posttreatment visit and remain clear during the 5 year follow-up period.

SECONDARY OUTCOMES:
To evaluate the safety and cosmetic outcome of once daily 5 days per week dosing for 6 weeks with imiquimod 5% cream in the treatment of sBCC

CONTACTS AND LOCATIONS:
Locations (1):
- Univertätsklinik für Dermatologie und Venerologie, Magedeburg, Germany